CLINICAL TRIAL: NCT02009891
Title: The Application of a Validated Patient and Clinic Specific Predictive Model to Reduce the Incidence of Multiple Births Resulting From Fresh In Vitro Fertilization Cycles
Brief Title: Use of Predictive Model to Assist Patients Having an Embryo Transfer After IVF
Status: Completed | Type: Observational
Sponsor: Ottawa Fertility Centre (Other)
Responsible Party: Principal Investigator, Dr. Arthur Leader, Consultant, Ottawa Fertility Centre
Other Study IDs: 100OFC
Record Dates: First submitted 2013-12-09; First posted 2013-12-12 (Estimated); Last update posted 2017-09-25 (Actual); Status verified 2017-09

CONDITIONS: Infertility
Keywords: predictive model; in vitro fertilization; elective single embryo transfer
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Control: Control couples who will not use predictive model
- Predictive model: Couples who will use predictive model

SUMMARY:
To determine in women undergoing IVF who are at high risk of multiple births (>35%), as calculated by the application of a predictive model - IVFsingleTM, if single embryo transfer will lead to both comparable clinical pregnancy rate (CPR) and other secondary outcomes such as live birth rate (LBR) and cumulative live birth rate (cLBR) in comparison to DET while reducing the incidence of multiple births (a secondary outcome measure).

ELIGIBILITY:
Inclusion Criteria:

Under 38 1st or second IVF attempt

-

Exclusion Criteria:

Over 37 years old donor egg third or greater IVF attempt cancellation in previous cycle for poor response successful pregnancy with IVF -

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women under age 38 undergoing 1st or 2nd IVF treatment who havae not had previous IVF pregancy nor cancelled IVF cycle for poor response.
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2012-06; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Clinical pregnancy rate at 8 -10 weeks gestational age | 36 months

SECONDARY OUTCOMES:
Multiple pregnancy rate | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Arthur Leader, MD, Principal Investigator — University of Ottawa
Locations (1):
- Ottawa Fertility Centre, Ottawa, Ontario, Canada

REFERENCES:
- See also: Related Info — http://www.conceive.ca